CLINICAL TRIAL: NCT03579277
Title: Comparison of Functional Outcomes and Morbidity of the Radial Forearm Versus the Ulnar Forearm Free Flap: A Prospective, Randomized Trial
Brief Title: Radial Forearm Versus the Ulnar Forearm Free Flap
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inadequate enrollment
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Joshua Adkinson, Chief of Hand Surgery, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1712593520
Record Dates: First submitted 2018-01-24; First posted 2018-07-06 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Free Tissue Flaps
Keywords: Radial Forearm Free Flap; Ulnar Forearm Free Flap; Free Tissue Transfer

STUDY DESIGN:
Intervention Model Description: Subjects are assigned to one of two treatment arms
Who Masked: Investigator
Masking Description: To the extend possible based on the nature of the study, subjects and researchers will be masked from the treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radial forearm free flap (Active Comparator): Subjects in this arm will receive a radial forearm free flap.
  Interventions: Procedure: Radial Forearm Free Flap
- Ulnar forearm free flap (Active Comparator): Subjects in this arm will receive an ulnar forearm free flap.
  Interventions: Procedure: Ulnar Forearm Free Flap

INTERVENTIONS:
Procedure: Radial Forearm Free Flap — Subjects in this arm will undergo a radial forearm free flap.
  Arms: Radial forearm free flap
Procedure: Ulnar Forearm Free Flap — Subjects in this arm will undergo an ulnar forearm free flap.
  Arms: Ulnar forearm free flap

SUMMARY:
This study evaluates donor site outcomes in patients receiving radial forearm free flap reconstruction versus ulnar forearm free flap reconstruction. Patients who meet criteria for forearm free flap reconstruction are randomized to receiving either radial forearm free flap or ulnar forearm free flap reconstruction.

DETAILED DESCRIPTION:
The radial forearm free flap and the ulnar forearm free flap are both well-described procedures used for free tissue transfer in reconstructive surgery. Although forearm free flaps are frequently performed, there is insufficient prospective data looking at the morbidity of the radial compared to ulnar forearm free flaps. The goal of this research study is to characterize the outcomes for each of these two flaps, and to determine if there is surgical equipoise, or if one flap is better than the other.

ELIGIBILITY:
Inclusion Criteria:

* Patients with planned forearm free flap reconstruction
* Patients who are deemed equal surgical candidates for radial forearm free flap and ulnar forearm free flap reconstruction
* Preoperative Allen's test completed and passed
* Patients have the capacity to complete the informed consent process

Exclusion Criteria:

* Patients that are not candidates for a forearm flap based on their physiology
* Clinically evident peripheral neuropathy (e.g., diabetic neuropathy, leprosy)
* Patients requiring concurrent forearm bone for reconstruction
* Child, prisoner, or other vulnerable group

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Average Grip Strength (lbs) in the operative hand and non-operative hand | up to 6 months
  Subjects' grip strength in their operative hand and non-operative hand, each measured as the maximum amount of force applied by the hand to a Jamar Dynometer in pounds.
Average Key Pinch Strength (lbs) in the operative hand and non-operative hand | up to 6 months
  Subjects' pinch strength in their operative hand and non-operative hand, each measured as the maximum amount of force applied with key pinch in pounds.
Average Physician and Patient Rating of Scar Appearance | up to 6 months
  Subject's and physician's reported assessment of scar appearance on a Likert scale up to 10.
Aggregated Brief Michigan Hand Questionnaire results (composite score) | up to 6 months
  Subjects' reported outcomes of hand function, as measured by the brief Michigan Hand Questionnaire survey results, on a scale up to 100.
Average Static Two Point Discrimination (mm) | up to 6 months
  Subjects' static two point discrimination threshold in their finger pads, palm, and dorsum of the hand, in the operative and non-operative extremity, each measured in millimeters.

SECONDARY OUTCOMES:
Number of patients with complete flap loss | up to 6 months
  Number of patients with complete flap loss as assessed by chart review.
Number of patients with partial flap loss | up to 6 months
  Number of patients with partial flap loss as assessed by chart review.
Number of patients reporting cold intolerance | up to 6 months
  Number of patients reporting cold intolerance in the operative and non-operative extremity as assessed by patient's response to questioning them about feeling cold intolerance.
Number of patients reporting neuropathy | up to 6 months
  Number of patients reporting cold intolerance as assessed by patient's response to questioning them about feeling neuropathy
Number of patients with postoperative hematoma at donor site | up to 6 months
  Number of patients with postoperative hematoma at donor site, as assessed by chart review.
Number of patients with postoperative cellulitis at donor site | up to 6 months
  Number of patients with postoperative cellulitis at donor site as assessed by chart review.
Number of patients with postoperative hematoma at recipient site | up to 6 months
  Number of patient with postoperative hematoma at recipient site, as assessed by chart review
Number of patient with postoperative infection at recipient site | up to 6 months
  Number of patient with postoperative infection at recipient site, as assessed by chart review.
Number of patients experiencing mortality | up to 6 months
  Number of patients experiencing mortality, as assessed by chart review.
Number of patients with donor site dehiscence | up to 6 months
  Number of patients with donor site dehiscence, as assessed by chart review
Number of patients with partial skin graft non-take | up to 6 months
  Number of patients with partial skin graft non-take, as assessed by chart review
Number of patients with complete skin graft non-take | up to 6 months
  Number of patients with complete skin graft non-take, as assessed by chart review

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Adkinson, M.D., Principal Investigator — Indiana University School of Medicine
Locations (1):
- Eskenazi Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided